CLINICAL TRIAL: NCT03973008
Title: Phase III, Randomized, Open-label Study of Adjuvant Chemotherapy Combined With Chemoradiotherapy Versus Adujvant Chemotherapy After Standard D2 Resection for Locally Advanced Proximal Gastric Adenocarcinoma
Brief Title: Adujvant CT+CRT vs Adujvant CT After D2 Resection for Locally Advanced Proximal Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-GA-CRT
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastric Adenocarcinoma; Adjuvant Radiotherapy
MeSH Terms: interventions — Chemoradiotherapy, Adjuvant; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adujvant CT+CRT (Experimental): Four to six weeks after D2 radical surgery, adjuvant chemotherapy was initiated with SOX regimen , repeated every three weeks, and adjuvant radiotherapy was started at the end of two cycles of adjuvant chemotherapy , with synchronous tegiol single drug chemotherapy. And the original SOX regimen was continued for 4 cycles after 3-4 weeks of radiotherapy.
  Interventions: Radiation: Adjuvant Chemoradiotherapy; Drug: Adjuvant Chemotherapy
- Adujvant CT (Active Comparator): The adjuvant chemotherapy was started 4-6 weeks after D2 radical operation. The SOX regimen was repeated every 3 weeks for 8 cycles.
  Interventions: Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Radiation: Adjuvant Chemoradiotherapy — DT 45Gy/25F/5W, using IMRT technology, synchronous tegio single drug chemotherapy
  Other Names: CRT
  Arms: Adujvant CT+CRT
Drug: Adjuvant Chemotherapy — Oxalis 130mg/m2 intravenous drip on day 1, tegio 80-120 mg daily, twice, half an hour after breakfast and dinner, for 14 consecutive days
  Other Names: CT

SUMMARY:
This study evaluates the addition of adjuvant chemoradiotherapy to adjuvant chemotherapy in the treatment of locally advanced proximal gastric adenocarcinoma after standard D2 radical resection.

DETAILED DESCRIPTION:
Because of its special anatomical structure, local recurrence rate of locally advanced proximal gastric adenocarcinoma is still high after radical operation.

As a local/regional therapy, radiotherapy combined with concurrent chemotherapy can kill local residual tumor cells and reduce the risk of local and regional recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary Participation and Written Signature of Informed Consent.
* Age 18-70, gender unlimited.
* Gross pathology confirmed that the tumor center was within 1 cm to 5 cm of the EGJ line. Histopathologically diagnosed as adenocarcinoma.
* No neoadjuvant therapy.
* Transabdominal standard D2 radical operation was performed and R0 resection was performed. Ascites cytology was negative.
* The pathological stages were IIB, IIIA, IIIB and IIIC.
* There was no intraperitoneal implantation and distant metastasis. CT should be routinely performed to evaluate the tumor bed before radiotherapy. Positron emission tomography (PET-CT) could be accepted to determine whether there was residual or distant metastasis.
* Physical condition score ECOG 0-1.
* No history of serious heart and lung diseases, abnormal hematological examination and immunodeficiency: hemoglobin (Hb) > 9 g/dL; white blood cell (WBC) > 3 x 109/L; neutrophil (ANC) > 1.5 x 109/L; platelet (Pt) > 100 x 109/L; bilirubin < 1.5 times the upper limit of normal value; glutathione transaminase (ALT) & alanine transaminase (AST) = 2.5 times the upper limit of normal value; serum creatinine < 1.5 times the normal value Upper limit.
* No other systemic tumors were found.
* Fertile men or women are willing to take contraceptive measures in the trial.
* The daily energy intake is more than 1500 kcal.

Exclusion Criteria:

* Those who had a history of malignant tumors (except skin basal cell carcinoma, thyroid papillary adenocarcinoma and cervical carcinoma in situ, who survived for more than 3 years after treatment).
* Patients with a history of neoadjuvant radiotherapy and chemotherapy before operation.
* Study participants who participated in other clinical trials within 30 days before treatment.
* Pregnancy, lactation or fertility without contraceptive measures.
* Drug addiction and other adverse drug addiction, long-term alcoholism and AIDS patients.
* Those with uncontrollable infections, seizures, or loss of self-awareness due to mental illness.
* Those with a history of severe allergy or specific constitution.
* Researchers believe that it is not appropriate to participate in this experiment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 year
  after primary treatment the patient survives without any signs or symptoms of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Jinwen Shen, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Shen J, Zhu X, Du Y, Zhu Y, Yu P, Yang L, Xu Z, Huang L, Zhang Y, Zhang Y, Liu L, Cheng X. Adjuvant SOX chemotherapy versus concurrent chemoradiotherapy after D2 radical resection of locally advanced esophagogastric junction (EGJ) adenocarcinoma: study protocol for a randomized phase III trial (ARTEG). Trials. 2021 Oct 30;22(1):753. doi: 10.1186/s13063-021-05617-7. PMID 34717717